CLINICAL TRIAL: NCT06328504
Title: Efficacy of Cashew Nut Protein Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cashew Protocol
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
Keywords: cashew; food allergy; immunotherapy; children
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cashew Immunotherapy (Experimental): Children with cashew allergy receiving OIT (OIT-oral immunotherapy).
  Interventions: Combination Product: Cashew immunotherapy
- Cashew avoidance (No Intervention): Children with cashew allergy not receiving OIT (OIT-oral immunotherapy).

INTERVENTIONS:
Combination Product: Cashew immunotherapy — Following the building-up phase (up to 60 weeks), patients will receive a daily low dose of cashew flour (1200 mg cashew protein) mixed with well-tolerated fruit mousse for 3 months (12 +/- 3 weeks).
  Arms: Cashew Immunotherapy

SUMMARY:
It is a randomized, single-center, controlled trial to evaluate the effectiveness of oral immunotherapy with cashew protein compared with standard treatment (elimination diet) in pediatric patients with cashew allergy.

DETAILED DESCRIPTION:
According to Polish data, in the population of children suspected of food allergy, cashew was the third nut found to be allergic, after peanut and hazelnut. Allergic reactions to nuts can be severe and life-threatening, making it challenging to avoid hidden sources of the allergen.

An effective and safe alternative to allergen avoidance strategies may be the use of oral specific immunotherapy.

In this study 39 children, aged 4 to 17 years with a diagnosis of IgE-dependent allergy to cashew, confirmed by an open oral provocation test (OFC; the first provocation before starting oral desensitization), will be randomly (2:1) assigned to two groups. The first group will be desensitized with a maintenance dose - 1200mg of cashew protein, while the second group - the control group - will be offered standard management - avoidance of cashew consumption.

Patients in the control group will be offered immunotherapy at the end of the study if its effectiveness is confirmed.

The desensitization procedure was planned in accordance with the guidelines for immunotherapy in food allergy of the European Academy of Allergology and Clinical Immunology.

The source of cashew protein is flour. The first dose of immunotherapy is given to patients in the intervention group in the hospital ward. The size of the initial dose depends on the symptom-triggering dose during the initial oral food provocation with cashew protein.

Every 2 weeks in the hospital setting, another higher dose of cashew protein will be given to the child. The requirement for increasing the dose of cashew is to achieve full tolerance of the previous dose. The maximum duration of this phase is 60 weeks.

After the maximum dose is tolerated, desensitization will continue for 12 weeks - the maintenance phase of desensitization.

The maintenance dose is 1200mg of cashew protein. The duration of the maintenance phase is 12 weeks (+/-3 weeks). After 12 weeks +/-3 weeks of maintenance dose, OFC and cashew protein tolerance assessment will be performed. Confirmation of complete cashew tolerance is the tolerance of a dose of 4043mg of cashew protein. Primary outcomes include the proportion of participants tolerating a single dose of 4043mg cashew protein during the final oral food challenge. Secondary outcomes assess adverse events, changes in immunological parameters, and the maximum tolerated doses of cashew protein in each group.

ELIGIBILITY:
Inclusion Criteria:

* age between 4 and 17 years,
* IgE (immunoglobulin E) -mediated cashew allergy confirmed with positive skin prick tests with cashew allergens (diameter of the wheal greater than 3mm) and/or specific IgE (immunoglobulin E) level greater than 0.35-kilo units of Allergen per liter (kUA/l),
* allergic reaction to cashew protein during oral food challenge (OFC),
* Signed Informed Consent by parent/legal guardian and patient aged >16 years old,
* Patient's and caregivers' cooperation with the researcher.

Exclusion Criteria:

* no confirmed allergy to cashew,
* negative provocation test with cashew,
* severe asthma,
* mild/moderate asthma poorly controlled: FEV1 (forced expiratory volume at one second) <80% (less than 5 perc), FEV1/FVC (forced expiratory volume at one second/forced vital capacity) <75% (less than 5 perc), hospitalization for asthma exacerbation in the past 12 months,
* oral/sublingual/subcutaneous immunotherapy to other allergens during the study,
* eosinophilic gastroenteritis,
* chronic diseases requiring ongoing treatment, including heart disease, epilepsy, metabolic diseases, diabetes,
* taking medications:

  * oral, daily steroid therapy >1 month in the past 12 months,
  * a minimum of 2 times oral steroid therapy (a period of at least 7 days) in the past 12 months,
  * one-time oral steroid therapy (min. 7 days) in the last 3 months,
  * biological treatment,
  * need to take antihistamines continuously,
  * therapy with β-blockers, ACE-inhibitors (angiotensin converting enzyme), calcium channel inhibitors,
* pregnancy,
* lack of consent to participate in the study,
* lack of patient cooperation.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2027-04-21 (Estimated)

PRIMARY OUTCOMES:
Cashew full tolerance | Up to 60 weeks of OIT (oral immunotherapy)
  Percentage of children tolerating a single dose of 4g of cashew protein after 12 weeks of immunotherapy at a maintenance dose.

SECONDARY OUTCOMES:
Cashew partial tolerance | Up to 60 weeks of OIT (oral immunotherapy)
  Percentage of children with partial tolerance, defined as an increase in the tolerated dose by at least 10-fold and tolerance of at least 1.2g of cashew protein but less than 4g of cashew protein at the end of 12 weeks of cashew protein immunotherapy at the maintenance dose or after 60 weeks of immunotherapy
OIT safety | Up to 60 weeks of OIT (oral immunotherapy)
  Number and type of side effects during oral desensitization with cashew protein, divided into mild, moderate and severe.
Wheal diameter in skin prick tests | Up to 60 weeks of OIT (oral immunotherapy)
  Difference in wheal diameter in skin prick tests between groups before and after completion of 12 weeks of cashew protein immunotherapy at the maintenance dose or after 60 weeks of immunotherapy.
SIgE (specific immunoglobulin E) (kUA/l) levels | Up to 60 weeks of OIT (oral immunotherapy)
  Difference in sIgE (specific immunoglobulin E) (kUA/l) levels against cashew, walnut, pistachio, peanut, hazelnut and almond allergens evaluated between groups 12 weeks of immunotherapy at maintenance dose or after 60 weeks of immunotherapy.
Basophil activation test (BAT) | Up to 60 weeks of OIT (oral immunotherapy)
  Difference in BAT test values between groups before and after 12 weeks of immunotherapy at maintenance dose or after 60 weeks of immunotherapy
Quality of life- FAQLQ (Food Allergy Quality of Life Questionnaire) | Up to 60 weeks of OIT (oral immunotherapy)
  Assessment of quality of life before and after desensitization (impact on families' lives) using FAQLQ. In children up to 12 years old we use FAQLQ-PF (Parent Form) and FAQLQ-CF (Child Form) in children 8-12 years old. For children 13-17 years old we use FAQLQ-TF (Teenager Form).
  These questionnaires are under validation in Polish and will be used if validation is completed.
  The FAQLQ-PF consists of 30 questions divided into three domains: Emotional Impact, Food Anxiety, and Social and Dietary Restrictions. Parents of children aged 4-6 years old answer 26 questions, and parents of children aged 7-12 years old answer all 30 questions. The FAIM (Food Allergy Independence Measure) consists of four questions and assesses parents expectations of their child's food allergy outcomes.
  FAQLQ- CF consist of 30 questions. FAQLQ- TF consist of 28 questions. Every question in all questionaires except FAIM part is assessed in 7 points scale, the higher value the worse outcome.
Air condensate | Up to 60 weeks of OIT (oral immunotherapy)
  Evaluation of pro-inflammatory cytokine levels in exhaled air condensate
IgG4 (immunoglobulin IgG4) (mgA/l) levels | Up to 60 weeks of OIT (oral immunotherapy)
  Difference in sIgG4 (immunoglobulin IgG4) (mgA/l) levels against cashew, walnut, pistachio, peanut, hazelnut and almond allergens evaluated between groups 12 weeks of immunotherapy at maintenance dose or after 60 weeks of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szczukocka-Zych, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393
- [Background] Bognanni A, Chu DK, Firmino RT, Arasi S, Waffenschmidt S, Agarwal A, Dziechciarz P, Horvath A, Jebai R, Mihara H, Roldan Y, Said M, Shamir R, Bozzola M, Bahna S, Fiocchi A, Waserman S, Schunemann HJ, Brozek JL; WAO DRACMA Guideline Group. World Allergy Organization (WAO) Diagnosis and Rationale for Action against Cow's Milk Allergy (DRACMA) guideline update - XIII - Oral immunotherapy for CMA - Systematic review. World Allergy Organ J. 2022 Sep 8;15(9):100682. doi: 10.1016/j.waojou.2022.100682. eCollection 2022 Sep. PMID 36185550
- [Background] de Silva D, Rodriguez Del Rio P, de Jong NW, Khaleva E, Singh C, Nowak-Wegrzyn A, Muraro A, Begin P, Pajno G, Fiocchi A, Sanchez A, Jones C, Nilsson C, Bindslev-Jensen C, Wong G, Sampson H, Beyer K, Marchisotto MJ, Fernandez Rivas M, Meyer R, Lau S, Nurmatov U, Roberts G; GA2LEN Food Allergy Guidelines Group. Allergen immunotherapy and/or biologicals for IgE-mediated food allergy: A systematic review and meta-analysis. Allergy. 2022 Jun;77(6):1852-1862. doi: 10.1111/all.15211. Epub 2022 Jan 19. PMID 35001400
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Bollinger ME, Dahlquist LM, Mudd K, Sonntag C, Dillinger L, McKenna K. The impact of food allergy on the daily activities of children and their families. Ann Allergy Asthma Immunol. 2006 Mar;96(3):415-21. doi: 10.1016/S1081-1206(10)60908-8. PMID 16597075
- [Background] Cox LS, Sanchez-Borges M, Lockey RF. World Allergy Organization Systemic Allergic Reaction Grading System: Is a Modification Needed? J Allergy Clin Immunol Pract. 2017 Jan-Feb;5(1):58-62.e5. doi: 10.1016/j.jaip.2016.11.009. PMID 28065342
- [Background] Anagnostou A. Food immunotherapy: current status and future needs. Expert Rev Clin Immunol. 2023 Jun;19(6):561-563. doi: 10.1080/1744666X.2023.2201438. Epub 2023 Apr 11. No abstract available. PMID 37038747
- [Background] Koplin JJ, Wake M, Dharmage SC, Matheson M, Tang ML, Gurrin LC, Dwyer T, Peters RL, Prescott S, Ponsonby AL, Lowe AJ, Allen KJ; HealthNuts study group. Cohort Profile: The HealthNuts Study: Population prevalence and environmental/genetic predictors of food allergy. Int J Epidemiol. 2015 Aug;44(4):1161-71. doi: 10.1093/ije/dyu261. Epub 2015 Jan 21. PMID 25613427
- [Background] Brough HA, Caubet JC, Mazon A, Haddad D, Bergmann MM, Wassenberg J, Panetta V, Gourgey R, Radulovic S, Nieto M, Santos AF, Nieto A, Lack G, Eigenmann PA. Defining challenge-proven coexistent nut and sesame seed allergy: A prospective multicenter European study. J Allergy Clin Immunol. 2020 Apr;145(4):1231-1239. doi: 10.1016/j.jaci.2019.09.036. Epub 2019 Dec 20. PMID 31866098
- [Background] Elizur A, Appel MY, Nachshon L, Levy MB, Epstein-Rigbi N, Koren Y, Holmqvist M, Porsch H, Lidholm J, Goldberg MR. Cashew oral immunotherapy for desensitizing cashew-pistachio allergy (NUT CRACKER study). Allergy. 2022 Jun;77(6):1863-1872. doi: 10.1111/all.15212. Epub 2022 Jan 15. PMID 35000223
- [Background] Chojnowska-Wojtowicz M, Lyzwa K, Zielinska J, Zagorska W, Grzela K. Prevalence of nut allergen sensitization among children in central Poland. Postepy Dermatol Alergol. 2023 Feb;40(1):40-46. doi: 10.5114/ada.2022.124730. Epub 2023 Feb 27. PMID 36909898
- [Background] Lyzwa K, Chojnowska-Wojtowicz M, Zielinska J, Zagorska W, Kulus M, Grzela K. Sensitization to nut allergens in children with food allergy and other atopic diseases - just a coexistence? Postepy Dermatol Alergol. 2023 Jun;40(3):402-410. doi: 10.5114/ada.2023.128991. Epub 2023 Jul 16. PMID 37545822
- [Derived] Szczukocka A, Pietrzyk-Kozinska M, Zielinska J, Krupa-Laska A, Krejner-Bienias A, Kulus M, Grzela K. Efficacy of cashew nut protein immunotherapy: protocol for a single-centre randomised controlled trial in a Polish paediatric population. BMJ Open. 2025 Jul 1;15(7):e101139. doi: 10.1136/bmjopen-2025-101139. PMID 40592755